CLINICAL TRIAL: NCT05022212
Title: Phase 2 Placebo-controlled Randomized Trial of LACTIN-V (Lactobacillus Crispatus CTV-05) Among Women at High Risk of HIV Acquisition in Durban, South Africa
Brief Title: Phase 2 Trial of LACTIN-V in Women at High Risk of HIV Acquisition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of KwaZulu (Other); Harvard University (Other); Aurum Institute (Other); Health Systems Trust (Other); Osel, Inc. (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LV-007; 1R01HD098978 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-08-26 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Bacterial Vaginosis; HIV Infections
Keywords: Vaginal microbiome; bacterial Vaginosis; HIV infections
MeSH Terms: conditions — Vaginosis, Bacterial; HIV Infections

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized, placebo-controlled trial of the vaginal live biotherapeutic product LACTIN-V in 60 young South African women, randomizing women 2:1 to LACTIN-V vs. placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LACTIN-V (Active Comparator): LACTIN-V contains a naturally occurring human vaginal strain of Lactobacillus (L.) crispatus CTV- 05. At a potency of 2 x 109 cfu/dose, it is preserved in powder formulation, and applied by a vaginal applicator.
  Women will receive the study product for five consecutive days, followed by twice weekly for three additional weeks. Women will be followed during the dosing (4 weeks) and post-dosing phase (4 weeks) for a total of 64 days.
  Interventions: Drug: LACTIN-V
- Placebo (Placebo Comparator): A matching placebo formulation without L. crispatus CTV-05 is supplied in an identical applicator containing just the powder formulation.
  Women will receive the placebo for five consecutive days, followed by twice weekly for three additional weeks. Women will be followed during the dosing (4 weeks) and post-dosing phase (4 weeks) for a total of 64 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LACTIN-V — administered vaginally
  Other Names: Lactobacillus crispatus CTV-05
  Arms: LACTIN-V
Drug: Placebo — administered vaginally
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the impact of LACTIN-V, a vaginally administered live biotherapeutic product (LBP) that contains the human L. crispatus CTV-05 strain, on the vaginal microbiome of Lactobacillus-deficient young women in the South African FRESH study who are at high risk for HIV acquisition.

DETAILED DESCRIPTION:
We will conduct a randomized, placebo-controlled trial of the vaginal live biotherapeutic product LACTIN-V in 60 young South African women.

After being informed about the study and potential risks, all participants giving written informed consent will be enrolled if they meet eligibility criteria. At enrollment on Day 1, they will start a 7-day course of standard oral metronidazole treatment for bacterial vaginosis. Women who completed their metronidazole treatment will be randomized 2:1 to LACTIN-V vs. placebo. Within 8-48 hours of the final metronidazole dose, women will receive the study product for five consecutive days, followed by twice weekly for three additional weeks. Women will be followed during the dosing (4 weeks) and post-dosing phase (4 weeks) for a total of 64 days.

ELIGIBILITY:
Inclusion Criteria:

1. FRESH study participant.
2. Capable of reading and writing English or isiZulu and voluntarily provide written informed consent to participate in the study and comply with all study procedures
3. HIV-negative
4. Nugent score 4-10 on vaginal Gram stain
5. Otherwise healthy women, 18-23 years of age on the day of enrolment
6. Regular predictable menstrual cycles or amenorrhoeic for at least 3 months due to use of a long-acting progestin.
7. Willing to complete 7-day course of oral metronidazole.
8. Willing to be asked questions about personal medical health and sexual history
9. Willing to apply study agent vaginally and comply with study examinations
10. Willing to self-administer Study Product on dosing days that do not coincide with regular FRESH study visits.
11. Agree to try to abstain from sexual intercourse 12 hours prior to study visits that include a gynaecological exam (Randomization Visit 3, Follow-up Visit 11, Final Visit 19).
12. Agree to try to abstain from sexual intercourse for 12 hours after study product administration to ensure that the product will remain inside the vagina.
13. Agree to abstain from the use of any other vaginal product throughout the trial period from the time of enrolment through the end of the study.

    Note: Intravaginal products include contraceptive creams such as Gynol II, gels, foams, sponges, lubricants not approved by the study investigators, tampons and douches.
14. Must be stable on a reliable method of long-acting birth control and agree to remain on, for the duration of the study (if of childbearing potential) or, of non-childbearing potential (permanently sterile).

Exclusion Criteria:

1. Urogenital infection (as tested during the FRESH Week 5 Study Visit, reported within 30 days of detection at the LACTIN-V Enrolment Visit).

   Note: Urogenital infection includes urinary tract infection, Trichomonas (T.) vaginalis, Neisseria (N.) gonorrhoeae, Chlamydia (C.) trachomatis, Mycoplasma genitalium.
2. Diagnosis of two or more outbreaks of N. gonorrhoeae, C. trachomatis, T. vaginalis, Mycoplasma genitalium, or herpes simplex virus (herpes genitalis) within 6 months prior to enrolment.
3. Subject is ineligible if menstrual cycle length is less than 21 days
4. Subject is ineligible if deep epithelial disruption is observed on genital examination noted on or before the Randomization Visit
5. Positive for HIV (as tested during the FRESH Week 5 Study Visit, within 30 days of the LACTIN-V Enrolment Visit).
6. Current pregnancy or within 2 months of last pregnancy
7. Vaginal or systemic antibiotic or antifungal therapy within 21 days of enrolment
8. Use of disulfiram within past 2 weeks or other contraindication to use of metronidazole
9. Any condition requiring regular periodic use of systemic antibiotics during participation in the trial
10. Investigational drug use other than LACTIN-V within 30 days or 10 half- lives of the drug, whichever is longer, of Enrolment Visit
11. Other planned participation in an investigational drug study while participating in this study
12. Intrauterine device (IUD) insertion or removal, pelvic surgery, cervical cryotherapy or cervical laser treatment within the last 2 months prior to enrolment
13. Use of vaginal ring (e.g, NuvaRing) within 3 days of enrolment or during the course of the study
14. Hysterectomy
15. Unwilling to complete 7 days of oral metronidazole (twice daily) with the last dose taken no later than 48 hours prior to randomization (minimum of 12 of 14 doses required)
16. Use of new long-acting hormonal treatments. Participant may be enrolled if stable (>1 month) on existing therapy as determined by the principal investigator (PI)
17. Known allergy to any component of LACTIN-V/placebo or metronidazole or to nitroimidazole derivatives or latex (condoms)
18. Any social, medical, or psychiatric condition including history of drug or alcohol abuse that in the opinion of the investigator would make it difficult for the participant to comply with study procedures
19. Any serious or chronic illness, deemed incompatible with study participation by the study doctor, including immunosuppression due to cancer chemotherapy, systemic corticosteroids.

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- FRESH (Females Rising through Education, Support and Health) Clinical Research Site, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosmann C, Anahtar MN, Handley SA, Farcasanu M, Abu-Ali G, Bowman BA, Padavattan N, Desai C, Droit L, Moodley A, Dong M, Chen Y, Ismail N, Ndung'u T, Ghebremichael MS, Wesemann DR, Mitchell C, Dong KL, Huttenhower C, Walker BD, Virgin HW, Kwon DS. Lactobacillus-Deficient Cervicovaginal Bacterial Communities Are Associated with Increased HIV Acquisition in Young South African Women. Immunity. 2017 Jan 17;46(1):29-37. doi: 10.1016/j.immuni.2016.12.013. Epub 2017 Jan 10. PMID 28087240
- [Background] Mitchell C, Manhart LE, Thomas K, Fiedler T, Fredricks DN, Marrazzo J. Behavioral predictors of colonization with Lactobacillus crispatus or Lactobacillus jensenii after treatment for bacterial vaginosis: a cohort study. Infect Dis Obstet Gynecol. 2012;2012:706540. doi: 10.1155/2012/706540. Epub 2012 May 30. PMID 22693410
- [Background] Cohen CR, Wierzbicki MR, French AL, Morris S, Newmann S, Reno H, Green L, Miller S, Powell J, Parks T, Hemmerling A. Randomized Trial of Lactin-V to Prevent Recurrence of Bacterial Vaginosis. N Engl J Med. 2020 May 14;382(20):1906-1915. doi: 10.1056/NEJMoa1915254. PMID 32402161
- [Background] Hemmerling A, Harrison W, Schroeder A, Park J, Korn A, Shiboski S, Cohen CR. Phase 1 dose-ranging safety trial of Lactobacillus crispatus CTV-05 for the prevention of bacterial vaginosis. Sex Transm Dis. 2009 Sep;36(9):564-9. doi: 10.1097/OLQ.0b013e3181a74924. PMID 19543144
- [Background] Hemmerling A, Harrison W, Schroeder A, Park J, Korn A, Shiboski S, Foster-Rosales A, Cohen CR. Phase 2a study assessing colonization efficiency, safety, and acceptability of Lactobacillus crispatus CTV-05 in women with bacterial vaginosis. Sex Transm Dis. 2010 Dec;37(12):745-50. doi: 10.1097/OLQ.0b013e3181e50026. PMID 20644497
- [Background] Cohen CR, Duerr A, Pruithithada N, Rugpao S, Hillier S, Garcia P, Nelson K. Bacterial vaginosis and HIV seroprevalence among female commercial sex workers in Chiang Mai, Thailand. AIDS. 1995 Sep;9(9):1093-7. doi: 10.1097/00002030-199509000-00017. PMID 8527084
- [Background] Mitchell C, Fredricks D, Agnew K, Hitti J. Hydrogen Peroxide-Producing Lactobacilli Are Associated With Lower Levels of Vaginal Interleukin-1beta, Independent of Bacterial Vaginosis. Sex Transm Dis. 2015 Jul;42(7):358-63. doi: 10.1097/OLQ.0000000000000298. PMID 26222747
- [Background] Ngugi BM, Hemmerling A, Bukusi EA, Kikuvi G, Gikunju J, Shiboski S, Fredricks DN, Cohen CR. Effects of bacterial vaginosis-associated bacteria and sexual intercourse on vaginal colonization with the probiotic Lactobacillus crispatus CTV-05. Sex Transm Dis. 2011 Nov;38(11):1020-7. doi: 10.1097/OLQ.0b013e3182267ac4. PMID 21992977
- [Derived] Hemmerling A, Govender V, Dong K, Dong M, Pillay S, Ndung'u T, Bhoola A, Moodley J, Casillas G, Lagenaur L, Mitchell CM, Kwon DS, Cohen CR. Acceptability of the live biotherapeutic LACTIN-V (Lactobacillus crispatus CTV-05) among young women at high risk of HIV acquisition in South Africa: data from the phase 2 placebo-controlled trial. Front Reprod Health. 2025 Mar 25;7:1544458. doi: 10.3389/frph.2025.1544458. eCollection 2025. PMID 40206350
- [Derived] Hemmerling A, Mitchell CM, Demby S, Ghebremichael M, Elsherbini J, Xu J, Xulu N, Shih J, Dong K, Govender V, Pillay V, Ismail N, Casillas G, Moodley J, Bergerat A, Brunner T, Liebenberg L, Ngcapu S, Mbano I, Lagenaur L, Parks TP, Ndung'u T, Kwon DS, Cohen CR. Effect of the vaginal live biotherapeutic LACTIN-V (Lactobacillus crispatus CTV-05) on vaginal microbiota and genital tract inflammation among women at high risk of HIV acquisition in South Africa: a phase 2, randomised, placebo-controlled trial. Lancet Microbe. 2025 Jun;6(6):101037. doi: 10.1016/j.lanmic.2024.101037. Epub 2025 Apr 4. PMID 40194532

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 were randomized to study product. 8 became then ineligible for randomization for the following reasons:
  * Not completing metronidazole course (n=1)
  * Acute UTI, STD, or vaginal infection besides BV (n=2)
  * Any condition requiring use of systemic antibiotics during the trial (n=2)
  * floods impacting on site access (n=2)
  * site disruption because of social unrest (n=1)
Groups:
- LACTIN-V: LACTIN-V contains a naturally occurring human vaginal strain of Lactobacillus (L.) crispatus CTV- 05. At a potency of 2 x 109 cfu/dose, it is preserved in powder formulation, and applied by a vaginal applicator.
  Women will receive the study product for five consecutive days, followed by twice weekly for three additional weeks. Women will be followed during the dosing (4 weeks) and post-dosing phase (4 weeks) for a total of 64 days.
  LACTIN-V: administered vaginally
- Placebo: A matching placebo formulation without L. crispatus CTV-05 is supplied in an identical applicator containing just the powder formulation.
  Women will receive the placebo for five consecutive days, followed by twice weekly for three additional weeks. Women will be followed during the dosing (4 weeks) and post-dosing phase (4 weeks) for a total of 64 days.
  Placebo: administered vaginally
Period: Overall Study
Arm/Group | LACTIN-V | Placebo
Started | 32 | 13
Completed | 32 | 11
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LACTIN-V | Placebo | Total
Number analyzed (Participants) | 32 | 13 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 13 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 13 | 45
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 13 | 45
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 32 | 13 | 45
Vaginal Gram Stain with Nugent Score 4-10 [Number; unit: participants] — The Nugent Score has values from 0 -10. 0-3 describes an optimal vaginal microbiome with lactobacilli but little bacterial diversity, 4-6 is an intermediate score, and 7-10 characterizes a vaginal microbiome with few lactobacilli and an overgrowth of pathogens.
  participants | 32 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Genital Tract Inflammation
Description: The proportion of participants with decreased genital tract proinflammatory cytokines and HIV target cells over 64 days of follow up, compared to levels at baseline.
  The outcome will be a change in immune parameters after treatment with LACTIN-V in comparison to placebo (proinflammatory cytokines in genital fluid, activated endocervical HIV target cells and the anti-HIV effect of vaginal secretions), measured as the number and proportions of endocervical CD4+ HIV target cells (i.e., CD4+/CCR5+/HLA-DR+/CD38+ T cells) at Day 64.
  Decreased inflammation will be defined using a measure of >1 log10 decrease in 3/8 markers between baseline and Day 64.
Time Frame: over 64 days
Population: Available samples at baseline and Day 64: LACTIN-V n=30, Placebo n=11. The comparison of the LACTIN-V vs. placebo arms was performed on a modified Intent to Treat (mITT) population, excluding one placebo participant who was erroneously dispensed two doses of LACTIN-V.
  Additionally, missing samples at Day 64 from two participants in the LACTIN-V group and one participant in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 30 | 11
Participants | 3 | 2

2. Primary Outcome: Number of Participants With Lactobacillus-dominant Vaginal Microbiota
Description: The proportion of participants with Lactobacillus-dominant vaginal microbiota in young South African women.
  Measured will be dominance of Lactobacillus crispatus (defined as > 50% relative abundance) after the intervention.
  Our primary outcome is measured at Day 36 (after 4 weeks of treatment with LACTIN-V), and at Day 64 (following the post- dosing phase).
Time Frame: over 64 days
Population: The comparison of the LACTIN-V vs. placebo arms was performed on a modified Intent to Treat (mITT) population, excluding one placebo participant who was erroneously dispensed two doses of LACTIN-V.
  Available samples at Day 36: LACTIN-V n=32, Placebo n=12. Available samples at Day 64: LACTIN-V n=31, Placebo n=11.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 32 | 12
Participants
  L. crispatus dominant vaginal bacterial community (> 50% relative abundance) on Day 36 | 13 | 0
  L. crispatus dominant vaginal bacterial community (> 50% relative abundance) on Day 64: number analyzed (Participants) | 31 | 11
  L. crispatus dominant vaginal bacterial community (> 50% relative abundance) on Day 64 | 8 | 1

3. Primary Outcome: Number of Participants With Vaginal Colonization of L. Crispatus CTV-05
Description: The proportion of participants experiencing successful colonization with L. crispatus CTV-05 following dose of study product through the final visit (Day 64) in the LACTIN-V arm.
  This primary outcome is measured at Day 36 (after 4 weeks of treatment with LACTIN-V), and at Day 64 (following the post- dosing phase).
Time Frame: over 64 days
Population: The comparison of the LACTIN-V vs. placebo arms was performed on a modified Intent to Treat (mITT) population, excluding one placebo participant who was erroneously dispensed two doses of LACTIN-V.
  Additionally, at Day 64 a missing sample from one participant in the placebo group.
  Available samples at Day 36: LACTIN-V n=32, Placebo n=12. Available samples at Day 64: LACTIN-V n=32, Placebo n=11.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 32 | 12
Participants
  Detection of L. crispatus CTV-05 at Day 36 | 22 | 1
  Detection of L. crispatus CTV-05 at Day 64: number analyzed (Participants) | 32 | 11
  Detection of L. crispatus CTV-05 at Day 64 | 15 | 1

4. Primary Outcome: Number of Participants With Vaginal Dysbiosis Indicated by a Nugent Score 4-10 on Vaginal Gram Stain
Description: The proportion of participants with a positive test for vaginal dysbiosis (Nugent Score 4-10 on vaginal Gram Stain) in each study arm by Day 36 and Day 64.
  The Nugent Score has values from 0 -10. 0-3 describes an optimal vaginal microbiome with lactobacilli but little bacterial diversity, 4-6 is an intermediate score, and 7-10 characterizes a vaginal microbiome with few lactobacilli and an overgrowth of pathogens.
Time Frame: over 64 days
Population: The comparison of the LACTIN-V vs. placebo arms was performed on a modified Intent to Treat (mITT) population, excluding one placebo participant who was erroneously dispensed two doses of LACTIN-V.
  Additionally, at Day 36 a missing sample from one participant in the LACTIN-V group.
  Available samples at Day 36: LACTIN-V n=31, Placebo n=12. Available samples at Day 64: LACTIN-V n=32, Placebo n=12.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 32 | 12
Participants
  Nugent Score 4-10 on Vaginal Gram Stain at Day 36: number analyzed (Participants) | 31 | 12
  Nugent Score 4-10 on Vaginal Gram Stain at Day 36 | 12 | 6
  Nugent Score 4-10 on Vaginal Gram Stain at Day 64 | 15 | 6

5. Primary Outcome: Number of Participants Reporting Any Solicited Adverse Events (AEs) Through the Final Visit
Description: Overall Safety of LACTIN-V and the applicator will be measured by the proportion of participants reporting any solicited Adverse Events (AEs) through the final visit on Day 64, compared between study arms.
Time Frame: over 64 days
Population: All 45 participants are included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 32 | 13
Participants | 26 | 9

6. Primary Outcome: Number of Participants Willing to Use This Type of Product in the Future
Description: Acceptability of LACTIN-V and the applicator will be measured by standardized questionnaire about acceptability of the study product and participants' stated willingness to use this type of product in the future, in each study arm. (Question "I would use the product again", on Day 36)
Time Frame: over 36 days
Population: Available acceptability data at Day 36: LACTIN-V n=30, Placebo n=13. Missing data from two participants in the LACTIN-V group.
Measure: Count of Participants; unit: Participants
Arm/Group | LACTIN-V | Placebo
Number analyzed (Participants) | 30 | 13
Participants
  strongly agree | 11 | 3
  agree | 11 | 7
  neutral | 5 | 3
  disagree | 2 | 0
  strongly disagree | 1 | 0

ADVERSE EVENTS:
Time Frame: 64 days
Arm/Group | LACTIN-V | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/13
Other Adverse Events (participants affected / at risk) | 26/32 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LACTIN-V (N=32) | Placebo (N=13)
Abnormal vaginal discharge (Reproductive system and breast disorders) | 9 | 2
Abnormal vaginal odor (Reproductive system and breast disorders) | 3 | 0
external genital irritiation (Reproductive system and breast disorders) | 1 | 0
external genital swelling (Reproductive system and breast disorders) | 1 | 0
genital itching or burning (Reproductive system and breast disorders) | 8 | 4
vaginal bleeding other than menstruation (Reproductive system and breast disorders) | 18 | 5
abdominal pain / cramps (Reproductive system and breast disorders) | 6 | 1
constipation (Gastrointestinal disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 1
frequent urination (Renal and urinary disorders) | 1 | 0
headache (Nervous system disorders) | 6 | 0
nausea (General disorders) | 2 | 0
pain/ burning with urination (Renal and urinary disorders) | 0 | 2
vomiting (General disorders) | 0 | 1
abnormal discharge (Reproductive system and breast disorders) | 2 | 0
urine odor (Renal and urinary disorders) | 1 | 0
toothache (Gastrointestinal disorders) | 1 | 0
pustule (Infections and infestations) | 1 | 0
folliculitis (Infections and infestations) | 1 | 0
chest discomfort (General disorders) | 1 | 0
eye infection, viral (Infections and infestations) | 1 | 0
viral skin infection (Infections and infestations) | 1 | 0
papular rash (Skin and subcutaneous tissue disorders) | 1 | 0 — papular pruritic fine erythematous left abdominal flank rash, deemed related to study product, study day 7-12
headache (Nervous system disorders) | 2 | 0
dizziness (Nervous system disorders) | 1 | 0
genital ulceration (Reproductive system and breast disorders) | 1 | 0 — clinical diagnosis as genital herpes ulceration
chlamydial infection (Infections and infestations) | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
subcutaneous abscess (Infections and infestations) | 1 | 0 — left axillary

LIMITATIONS AND CAVEATS:
In consideration of a set of circumstances that complicated the study progress (a 1-year delay of study start because of COVID-19 in 2020, a further 4-month delay because of destruction of the clinic site during social unrest in July 2021, and expiration of study product in March 2023), the study team together with the DSMB and the sponsor NICHD decided to stop enrollment at the end of 2022 at n=45, instead of the initial goal of n=60.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT05022212/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT05022212/ICF_001.pdf